CLINICAL TRIAL: NCT03295253
Title: Evaluation of Fat Grafting Technique Using Autologous Micro-fragmented Autologous Adipose Tissue Lipogems in Female Patients Suffering From Stress Urinary Incontinence
Brief Title: Fat Grafting Technique Using Autologous Adipose Tissue Lipogems in Patients Suffering From Stress Urinary Incontinence
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Miriam Hospital (Other)
Responsible Party: Principal Investigator, Janice Santos Cortes, Assistant Professor of Surgery (Urology), The Miriam Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 212516
Record Dates: First submitted 2017-08-02; First posted 2017-09-27 (Actual); Last update posted 2017-09-27 (Actual); Status verified 2017-09

CONDITIONS: Urinary Incontinence,Stress
Keywords: urinary incontinence; stress urinary incontinence; stress incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress; Urinary Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Female patients with Stress Incontinence (Experimental): Female patients who will undergo autologous adipose tissue harvesting/grafting using Lipogems and grafting in urethra/bladder neck
  Interventions: Procedure: Autologous adipose tissue harvesting/grafting using Lipogems

INTERVENTIONS:
Procedure: Autologous adipose tissue harvesting/grafting using Lipogems — Adipose tissue harvesting and grafting in the urethra using fat micro-fragmentation and processing device Lipogems

SUMMARY:
Urinary incontinence affects more than 200 million people worldwide. In women, childbirth or menopausal aging atrophic vagina, lack of estrogen stimulation of muscular turgor of the vagina, decrease tone of the urogenital diaphragm, attenuation and weakening of the urethral sphincter all result in stress incontinence, urge incontinence and sometimes mixed incontinence respectively.

The purpose of this study is to evaluate reconstructive lipoplasty with micro-fragmented autologous adipose tissue (Lipogems®) in female patients with stress urinary incontinence. This is a prospective study of 25 subjects that will be evaluated over a period of one year.

The treatment consist of the injection of micro fragmented adipose tissue, previously extracted from the patient in the area of the urethral sphyncter.

Patients will have follow ups at 6 months with Urodynamic studies to measure the pre-post injection differences to-date. Visual analog score questionnaire and report in subjective improvement, pad use and stress cough test will be documented at 1, 3, 6, and 12 months follow-up.

DETAILED DESCRIPTION:
Urinary incontinence affects more than 200 million people worldwide. In women, childbirth or menopausal aging atrophic vagina, lack of estrogen stimulation of muscular turgor of the vagina, decrease tone of the urogenital diaphragm, attenuation and weakening of the urethral sphincter all result in stress incontinence, urge incontinence and sometimes mixed incontinence respectively. The purpose of this study is to evaluate reconstructive lipoplasty with micro-fragmented autologous adipose tissue (Lipogems®) in female patients with stress urinary incontinence. This is a prospective study of 25 subjects that will be evaluated over a period of one year.

Different available treatments for stress urinary incontinence (SUI) are surgical: MMK, R A Z, Burch, (TOT, T VT-mesh sling) and urethral bulking agents. New treatments using mesenchymal stem cells have been tested for the last eight years and now moved from animal models to humans with positive results.

Subjects will receive a full history and examination by a single urologist. A clear history of their incontinence pattern, the amount of incontinence based on PAD counts, under what conditions incontinence occurs to categorize type of incontinence for the female patient pre- or post-menopause. Childbirth history, age of onset, time of occurrence, predisposing factors, medications, hormones, etc. all patients will be registered and categorized according to incontinence.

The patients will receive reconstructive lipoplasty with micro-fragmented autologous adipose tissue (Lipogems®).

Subjects will log their results immediately post injection and then daily for up to two years noting any changes they've noticed in their presenting problems. At 6 months Urodynamic studies will be performed to measure the pre-post injection differences to-date. Visual analog score questionnaire and report in subjective improvement, pad use and stress cough test will be documented at 1, 3, 6, and 12 months follow-up.

ELIGIBILITY:
Inclusion Criteria:

Female patients with:

1. stress incontinence (SUI)
2. mixed urinary incontinence (SUI main component)
3. Intrinsic Sphincter Deficiency (ISD)

Exclusion Criteria:

1. Present diagnosis of cancer (not in remission)
2. Patients with uncorrected vaginal prolapse (cystocele or utero/bladder prolapse)
3. Incontinence of unknown etiology (other medical reasons) overflow incontinence
4. Patients with neurogenic bladder
5. Any patients unable to give informed consent, including members of vulnerable populations
6. Patients with concomitant pelvic floor disorders, like interstitial cystitis or pelvic floor dysfunction
7. Vulvar dermatosis, herpes simplex or active or recurrent urinary tract infection
8. Patients with chronic steroid use
9. Patients 17 and under

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2016-12-15 (Actual); Primary Completion 2018-12-15 (Estimated); Study Completion 2018-12-15 (Estimated)

PRIMARY OUTCOMES:
Resolution of Stress urinary Incontinence Measured by patient reported outcomes on questionnaire | 2 years
  Comparison of pre and post procedure patient reported outcomes questionnaire
Resolution of Stress urinary Incontinence Measured by patient outcomes on Urodynamic Studies | 2 years
  Comparison of pre and post procedure patient Urodynamic studies
Resolution of Stress urinary Incontinence Measured by patient reported pad count | 2 years
  Comparison of pre and post procedure patient pad count
Resolution of Stress urinary Incontinence Measured by patient cough stress test | 2 years
  Comparison of pre and post procedure patient cough stress test

OTHER OUTCOMES:
Incidence of treatment related adverse events | 2 years
  site-reported adverse events designated as related to the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Janice Santos, MD, Principal Investigator — Women Medicine Collaborative/The Miriam Hospital; Patrizia Curran, MD, Study Director — The Miriam Hospital/ Women Medicine Collaborative
Locations (1):
- The Miriam Hospital/ Women Medicine Collaborative, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No